CLINICAL TRIAL: NCT02559271
Title: Pediatric Refraction With SVOne Autorefractor
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Smart Vision Labs (Industry)
Collaborators: State University of New York College of Optometry (Other)
Responsible Party: Sponsor
Other Study IDs: Aug/25/2015
Record Dates: First submitted 2015-09-21; First posted 2015-09-24 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-09

CONDITIONS: Ocular Refraction

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The study is used to verify the accuracy and repeatability of Smart Vision Labs Refractor in a pediatric population (between 5 and 16 years of age).

ELIGIBILITY:
Inclusion Criteria:

1. healthy children
2. ages 5-16 year
3. male and female

Exclusion Criteria:

1. presence of ocular disease
2. refractive surgery
3. amblyopia

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: pediatric population, between 5 and 16 years of age
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2015-08; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Sphere refraction measurement | up to 6 months
  the outcome include sphere refraction (in diopter) measurements by using both Smart Vision Labs autorefractor and subjective refraction
Cylinder refraction measurement | up to 6 months
  the outcome include cylinder refraction (in diopter) measurements by using both Smart Vision Labs autorefractor and subjective refraction
difference between two Sphere refraction measurements on the same patient | up to 6 months
  the outcome include the difference (in diopter) between two Sphere refraction measurements on the same patient by using smart vision labs autorefractor
difference between two cylinder refraction measurements on the same patient | up to 6 months
  the outcome include the difference (in diopter) between two cylinder refraction measurements on the same patient by using smart vision labs autorefractor

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Ciuffreda, PH.D, Principal Investigator — State University of New York College of Optometry
Locations (1):
- SUNY/College of Optometry, New York, New York, United States